CLINICAL TRIAL: NCT00111319
Title: An Open-Label, Randomized Study of VELCADE/Melphalan/Prednisone Versus Melphalan/Prednisone in Subjects With Previously Untreated Multiple Myeloma
Brief Title: VELCADE/Melphalan/Prednisone Versus Melphalan/Prednisone in Patients With Previously Untreated Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Clinical Research Monitor, Millennium Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-MMY-3002; NCT00109902 (obsolete NCT alias)
Expanded Access: Available
Record Dates: First submitted 2005-05-19; First posted 2005-05-20 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Multiple Myeloma
Keywords: Front Line; Multiple Myeloma; Untreated
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
The primary reason for this study is to determine whether the addition of VELCADE (bortezomib) for injection to standard melphalan/prednisone (MP) therapy improves the time to disease progression (TTP) in subjects with previously untreated multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

* Male or female
* Not a candidate for HDT/SCT due to: age - subject is 65 years or older or in subjects less than 65 years of age - presence of important comorbid condition(s) likely to have a negative impact on tolerability of HDT/SCT.
* Symptomatic multiple myeloma or asymptomatic multiple myeloma with related organ or tissue damage. Asymptomatic multiple myeloma-related organ or tissue damage can include presence of asymptomatic lytic bone lesion or plasmacytoma, or presence of anemia, renal function impairment, or hypercalcemia, as long as the criteria for pre-treatment clinical laboratory values indicated below are met.
* Presence of measurable disease, defined as:

  * For secretory multiple myeloma, measurable disease is defined as any quantifiable serum monoclonal protein value.
  * For oligosecretory or nonsecretory multiple myeloma, measurable disease is defined by the presence of measurable soft tissue or organ (not bone) plasmacytomas as determined by clinical examination or applicable radiographs.
* Karnofsky performance status score of equal or greater then 60%.
* Willing and able to complete the PRO instruments
* Agrees to use an acceptable barrier method for contraception for the duration of the study (for male subjects); If female subjects are still having menstrual periods and are not surgically sterile, they must be practicing an effective method of birth control before entry, and throughout the study, and have a negative serum B-HCG pregnancy test at screening.
* Have pretreatment clinical laboratory values meeting the criteria as described in the protocol within 14 days before randomization.
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

* Diagnosis of smoldering multiple myeloma or monoclonal gammopathy of undetermined significance (MGUS, hypercalcemia, and renal insufficiency related to the monoclonal protein; and (if determined) proportion of plasma cells in the bone marrow of 10% or less.
* Diagnosis of Waldenström's disease or other conditions in which IgM M protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions
* Prior or current systemic therapy for multiple myeloma including steroids (with the exception of emergency use of a short course [maximum of 4 days] of steroids before randomization or of prior or current use of bisphosphonates)
* Radiation therapy within 30 days before randomization
* Plasmapheresis within 30 days before randomization
* Major surgery within 30 days before randomization (kyphoplasty is not considered major surgery)
* History of allergic reaction attributable to compounds containing boron or mannitol
* Peripheral neuropathy or neuropathic pain Grade 2 or higher.
* Uncontrolled or severe cardiovascular disease, including myocardial infarction, within 6 months of enrollment, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis
* Other malignancy within the past 5 years. Exceptions if treated and not active include the following: basal cell or nonmetastatic squamous cell carcinoma of the skin, cervical carcinoma in situ or International Federation of Gynecology and Obstetrics (FIGO) Stage 1 carcinoma of the cervix
* Concurrent medical condition or disease (e.g., active systemic infection, uncontrolled diabetes) that is likely to interfere with study procedures or results, or that, in the opinion of the investigator would constitute a hazard for participating in this study
* Use of any investigational drugs within 30 days before randomization
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, or family members of the employees or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Time to progression

SECONDARY OUTCOMES:
Progression-free survival, overall response rate, overall survival, time to first response, duration of response, CR rate, and patient reported outcomes as assessed using the EORTC QLQ-C30, FACIT-F and EQ-5D instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Mateos MV, Oriol A, Martinez-Lopez J, Teruel AI, Bengoechea E, Palomera L, de Arriba F, Esseltine DL, Cakana A, Pei L, van de Velde H, Miguel JS. Outcomes with two different schedules of bortezomib, melphalan, and prednisone (VMP) for previously untreated multiple myeloma: matched pair analysis using long-term follow-up data from the phase 3 VISTA and PETHEMA/GEM05 trials. Ann Hematol. 2016 Dec;95(12):2033-2041. doi: 10.1007/s00277-016-2835-3. Epub 2016 Oct 14. PMID 27738789
- [Derived] San Miguel JF, Schlag R, Khuageva NK, Dimopoulos MA, Shpilberg O, Kropff M, Spicka I, Petrucci MT, Palumbo A, Samoilova OS, Dmoszynska A, Abdulkadyrov KM, Delforge M, Jiang B, Mateos MV, Anderson KC, Esseltine DL, Liu K, Deraedt W, Cakana A, van de Velde H, Richardson PG. Persistent overall survival benefit and no increased risk of second malignancies with bortezomib-melphalan-prednisone versus melphalan-prednisone in patients with previously untreated multiple myeloma. J Clin Oncol. 2013 Feb 1;31(4):448-55. doi: 10.1200/JCO.2012.41.6180. Epub 2012 Dec 10. PMID 23233713
- [Derived] Delforge M, Dhawan R, Robinson D Jr, Meunier J, Regnault A, Esseltine DL, Cakana A, van de Velde H, Richardson PG, San Miguel JF. Health-related quality of life in elderly, newly diagnosed multiple myeloma patients treated with VMP vs. MP: results from the VISTA trial. Eur J Haematol. 2012 Jul;89(1):16-27. doi: 10.1111/j.1600-0609.2012.01788.x. Epub 2012 May 7. PMID 22469559
- [Derived] Rowen D, Brazier J, Young T, Gaugris S, Craig BM, King MT, Velikova G. Deriving a preference-based measure for cancer using the EORTC QLQ-C30. Value Health. 2011 Jul-Aug;14(5):721-31. doi: 10.1016/j.jval.2011.01.004. PMID 21839411
- [Derived] Dimopoulos MA, Mateos MV, Richardson PG, Schlag R, Khuageva NK, Shpilberg O, Kropff M, Spicka I, Palumbo A, Wu KL, Esseltine DL, Liu K, Deraedt W, Cakana A, Van De Velde H, San Miguel JF. Risk factors for, and reversibility of, peripheral neuropathy associated with bortezomib-melphalan-prednisone in newly diagnosed patients with multiple myeloma: subanalysis of the phase 3 VISTA study. Eur J Haematol. 2011 Jan;86(1):23-31. doi: 10.1111/j.1600-0609.2010.01533.x. Epub 2010 Nov 15. PMID 20874823
- [Derived] Harousseau JL, Palumbo A, Richardson PG, Schlag R, Dimopoulos MA, Shpilberg O, Kropff M, Kentos A, Cavo M, Golenkov A, Komarnicki M, Mateos MV, Esseltine DL, Cakana A, Liu K, Deraedt W, van de Velde H, San Miguel JF. Superior outcomes associated with complete response in newly diagnosed multiple myeloma patients treated with nonintensive therapy: analysis of the phase 3 VISTA study of bortezomib plus melphalan-prednisone versus melphalan-prednisone. Blood. 2010 Nov 11;116(19):3743-50. doi: 10.1182/blood-2010-03-275800. Epub 2010 Jul 13. PMID 20628153
- [Derived] San Miguel JF, Schlag R, Khuageva NK, Dimopoulos MA, Shpilberg O, Kropff M, Spicka I, Petrucci MT, Palumbo A, Samoilova OS, Dmoszynska A, Abdulkadyrov KM, Schots R, Jiang B, Mateos MV, Anderson KC, Esseltine DL, Liu K, Cakana A, van de Velde H, Richardson PG; VISTA Trial Investigators. Bortezomib plus melphalan and prednisone for initial treatment of multiple myeloma. N Engl J Med. 2008 Aug 28;359(9):906-17. doi: 10.1056/NEJMoa0801479. PMID 18753647